CLINICAL TRIAL: NCT06429124
Title: Time-Restricted Eating in Alzheimer's Disease : The T.R.E.A.D Trial
Brief Title: Time Restricted Eating in Alzheimer's Disease
Acronym: TREAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Arizona State University (Other); Karlsruhe Institute of Technology (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HX-23-500-347-30-03
Record Dates: First submitted 2024-04-29; First posted 2024-05-24 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Alzheimer's Disease; Mild Cognitive Impairment; Intermittent Fasting; Nutritional Strategies; Time Restricted Eating
MeSH Terms: conditions — Cognitive Dysfunction; Intermittent Fasting | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: We will execute the specific aims using a pre-post non-randomized study design in which all participants receive the intervention. Outcome assessments for specific aim 2 will include neuropsychological tests, blood biomarkers, and psychological well-being measured at baseline and after 3 months of intervention.
Masking Description: This study will not use any masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Participants will be instructed to follow a 16/8 regimen characterized by 16 hours of fasting and an 8-hour eating window daily, on approximately 5 days/week, for 3 months. Previous research has shown that 16 hours of fasting is feasible, safe and well-tolerated among older adults, and that most persons report easy adjustment (Anton, Lee et al. 2019, Lee, Sypniewski et al. 2020). The intervention will be implemented through individual and group sessions with participants and will involve extensive education, coaching, guidance, and support throughout the 3-month intervention. Educational materials on lifestyle factors including physical activity will be provided to each participant. We will be also be collecting data on physical activity and sedentary behavior. These data will be co-variates when we conduct the statistical analysis.
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — Participants will be instructed to follow a 16/8 regimen characterized by 16 hours of fasting and an 8-hour eating window daily, on approximately 5 days/week, for 3 months. Previous research has shown that 16 hours of fasting is feasible, safe and well-tolerated among older adults, and that most persons report easy adjustment (Anton, Lee et al. 2019, Lee, Sypniewski et al. 2020). The intervention will be implemented through individual and group sessions with participants and will involve extensive education, coaching, guidance, and support throughout the 3-month intervention. Educational materials on lifestyle factors including physical activity will be provided to each participant. We will be also be collecting data on physical activity and sedentary behavior. These data will be co-variates when we conduct the statistical analysis.

SUMMARY:
This pilot and feasibility study will enable the research team to determine the feasibility of implementing a time-restricted eating regimen among adults with mild cognitive impairment (MCI) and the impact of time-restricted eating on cognitive performance and biomarkers of metabolic health in this population. Study staff will execute the specific aims using a pre-post, non-randomized study design in which all participants receive the intervention. The intervention is a 16/8 time-restricted eating regimen characterized by fasting for 16 hours and eating within an 8-hour window on 5 days per week for 3 months. Assessments will be performed at baseline and after the 3-month time-restricted eating intervention with the following outcome measures.

Outcome measures for feasibility include participant recruitment, retention and metrics of acceptability, safety, and adherence to the intervention. Outcome measures for cognitive performance and metabolic health include neuropsychological tests, blood biomarkers, and surveys of psychological well-being.

DETAILED DESCRIPTION:
The goal of this pilot study on time restricted eating regimens in the mild cognitive impairment (MCI) patient population will be to determine the feasibility of implementing the intervention and impact of time-restricted eating on cognitive performance and biomarkers of metabolic health. Researchers at the Barrow Neurological Institute, Alzheimer's Disease Program in collaboration with the Arizona State University College of Health Solutions will execute the specific aims using a pre-post non-randomized study design in which all participants receive the intervention. Outcome assessments for specific aim 2 will include neuropsychological tests, blood biomarkers, and psychological well-being measured at baseline and after 3 months of intervention.

Participants will be instructed to follow a 16/8 regimen characterized by 16 hours of fasting and an 8-hour eating window daily, on approximately 5 days/week, for 3 months. Primary outcomes will include participant recruitment, retention, acceptability, safety, and adherence to the 16 hours of fasting and 8-hour eating window. Researchers hypothesize that participants who follow a time-restricted eating pattern will have improvements in attention, working memory and semantic fluency domains. Study staff hypothesize that there will be improvements or trends toward improvements in inflammatory and cardiometabolic biomarkers (i.e., interleukin-6, tumor necrosis factor alpha, C-reactive protein, insulin, hemoglobin A1c, and lipids).

The results of this project will provide critical preliminary data for a longer-term, large-scale, randomized controlled trial of time-restricted eating on cognitive trajectory among adults with MCI. The novel findings from the proposed project and future studies will contribute significantly to the body of knowledge that will advance the field, with the ultimate goal of preventing or delaying the progression of MCI to dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female outpatients 55-89 years of age.
2. Meet Mayo Clinic Criteria for MCI.
3. If taking medications that may affect one or more study outcome measures(such as donepezil and memantine),the participant must be on a stable dose for at least the preceding 3 months.
4. A body mass index ≥18.5 and <40.0 kg/m2.
5. Access to the internet through computer or smartphone.
6. Must have a collateral informant/study partner(e.g. spouse or adult child) who has significant direct contact with the patient and who is willing to accompany the patient to specified clinic visits and be available for telephone visits/Interviews.
7. An education level > 8 years.
8. A proficiency in speaking and reading English or having a family member who is proficient in reading and speaking English and is willing to serve as a translator.
9. Vision and hearing must be sufficient to comply with study procedures.

Exclusion Criteria:

1. Diabetes mellitus that requires insulin treatment or is not well managed.
2. An eating disorder.
3. A contraindication to time-restricted eating.
4. Daily eating window <11 hours/day on ≥3 days/week.
5. MMSE score ≤9 or patients diagnosed with severe dementia by a clinician.
6. In the opinion of the investigator, participation would not be in the best interest of the subject.
7. Taking prescription medications twice a day that need to be taken with food.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  Insulin resistance will be estimated using HOMA-IR.
Average number of days per week of time-restricted eating | The eating window is assessed daily throughout the 3-month intervention.
  Feasibility will be assessed based on the average number of days per week that participants eat within the 8-hour eating window. The intervention goal is 5 or more days per week.

SECONDARY OUTCOMES:
Physical Activity and Sedentary Behavior Questionnaire Score | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Physical Activity and Sedentary Behavior Questionnaire will assess active time and time spent on exercise (PASB-Q; English Version) (Sattler et al., 2020)
Memory as measured by the Comprehensive TrailMaking Test (CTMT) | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Comprehensive Trail Making Test (CTMT) is a measure of organized visual search, attention, set shifting and divided attention (Reynolds 2002).
Cognitive Impairment as measured by the Mini Mental State Examination (MMSE) | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Mini Mental State Examination (MMSE) is used extensively in clinical and research settings to systematically measure and assess mental status. It is an 11- question measure that tests five areas of cognitive function: orientation, registration, attention, and calculation, recall, and language (Folstein et al., 1975).
Verbal Memory as Measured by the Auditory VerbalLearning Test (AVLT) | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Auditory Verbal Learning Test (AVLT) evaluates verbal memory by presenting a 15- word list five times followed by attempted recall. This is followed by a second 15-word recall interference list, followed by recall of the original list (Rey A. 1964).
Working Memory as measured by the WAIS-IV Digit Span Forward/Backward | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Digit Span Forward/Backward is a subset of the Wechsler Adult Intelligence Scale (WAIS) that captures attention efficiency and working memory.
Psychological Flexibility as Measured by the Comprehensive Assessment of Acceptance and Commitment Therapy Process (CompACT) | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Comprehensive Assessment of Acceptance and Commitment Therapy Process (CompACT) is a 23 item questionnaire that measures ACT processes, including psychological flexibility (Francis et al., 2016).
Brief Resilience Scale (BRS) Score | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Brief Resilience Scale (BRS) has 6 items and is a reliable means of assessing resilience as the ability to bounce back or recover from stress (Smith et al., 2008).
Perceived Stress Scale (PSS) Score | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Perceived Stress Scale (PSS) is used for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. The scale also includes questions about current levels of experienced stress (Cohen et al, 1983).
Pittsburgh Sleep Quality Index (PSQI) Score | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire designed to measure sleep quality and disturbance over past month (Buysse et al.,1989).
WHO Quality of Life Questionnaire | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  The WHO QOL has four domains (physical health, psychological, social relationships, and environment). The four domain scores denote an individual's perception of quality of life in each particular domain (WHOQOL Group, 1998).
Hemoglobin A1c | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention)
  Glycemic control will be assessed by hemoglobin A1c obtained via venipuncture.
C-reactive protein | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  Levels of inflammatory biomarkers will be assessed by C-reactive protein obtained via venipuncture.
Blood Pressure | Will be assessed at baseline (pre-intervention) and after the 3-month intervention (post-intervention).
  Study staff will be obtaining a participant blood pressure using an electronic blood pressure cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Yonas E Geda, MD, MSc, Principal Investigator — Barrow Neurological Institute, Alzheimer's Disease and Cognitive Disorders Division
Locations (2):
- United States (2):
  - Arizona State University, College of Health Solutions, Phoenix, Arizona
  - Barrow Neurological Institute, Division of Alzheimer's Disease, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No
The results of this proposed Barrow Neurological Foundation project will provide critical preliminary data for a future large-scale R01 grant application to the National Institutes of Health (NIH), but no individual participant data will be shared.

REFERENCES:
- [Background] Anson RM, Guo Z, de Cabo R, Iyun T, Rios M, Hagepanos A, Ingram DK, Lane MA, Mattson MP. Intermittent fasting dissociates beneficial effects of dietary restriction on glucose metabolism and neuronal resistance to injury from calorie intake. Proc Natl Acad Sci U S A. 2003 May 13;100(10):6216-20. doi: 10.1073/pnas.1035720100. Epub 2003 Apr 30. PMID 12724520
- [Background] Anton SD, Lee SA, Donahoo WT, McLaren C, Manini T, Leeuwenburgh C, Pahor M. The Effects of Time Restricted Feeding on Overweight, Older Adults: A Pilot Study. Nutrients. 2019 Jun 30;11(7):1500. doi: 10.3390/nu11071500. PMID 31262054
- [Background] Anton SD, Moehl K, Donahoo WT, Marosi K, Lee SA, Mainous AG 3rd, Leeuwenburgh C, Mattson MP. Flipping the Metabolic Switch: Understanding and Applying the Health Benefits of Fasting. Obesity (Silver Spring). 2018 Feb;26(2):254-268. doi: 10.1002/oby.22065. Epub 2017 Oct 31. PMID 29086496
- [Background] Brookmeyer R, Gray S, Kawas C. Projections of Alzheimer's disease in the United States and the public health impact of delaying disease onset. Am J Public Health. 1998 Sep;88(9):1337-42. doi: 10.2105/ajph.88.9.1337. PMID 9736873
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Carlson AJ, Hoelzel F. Apparent prolongation of the life span of rats by intermittent fasting. J Nutr. 1946 Mar;31:363-75. doi: 10.1093/jn/31.3.363. No abstract available. PMID 21021020
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Dimitratos SM, German JB, Schaefer SE. Wearable Technology to Quantify the Nutritional Intake of Adults: Validation Study. JMIR Mhealth Uhealth. 2020 Jul 22;8(7):e16405. doi: 10.2196/16405. PMID 32706729
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Francis, A. W., D. L. Dawson and N. Golijani-Moghaddam (2016).
- [Background] Goodrick CL, Ingram DK, Reynolds MA, Freeman JR, Cider N. Effects of intermittent feeding upon body weight and lifespan in inbred mice: interaction of genotype and age. Mech Ageing Dev. 1990 Jul;55(1):69-87. doi: 10.1016/0047-6374(90)90107-q. PMID 2402168
- [Background] Goodrick CL, Ingram DK, Reynolds MA, Freeman JR, Cider NL. Differential effects of intermittent feeding and voluntary exercise on body weight and lifespan in adult rats. J Gerontol. 1983 Jan;38(1):36-45. doi: 10.1093/geronj/38.1.36. PMID 6848584
- [Background] Gudden J, Arias Vasquez A, Bloemendaal M. The Effects of Intermittent Fasting on Brain and Cognitive Function. Nutrients. 2021 Sep 10;13(9):3166. doi: 10.3390/nu13093166. PMID 34579042
- [Background] Halagappa VK, Guo Z, Pearson M, Matsuoka Y, Cutler RG, Laferla FM, Mattson MP. Intermittent fasting and caloric restriction ameliorate age-related behavioral deficits in the triple-transgenic mouse model of Alzheimer's disease. Neurobiol Dis. 2007 Apr;26(1):212-20. doi: 10.1016/j.nbd.2006.12.019. Epub 2007 Jan 13. PMID 17306982
- [Background] HARMAN D. Aging: a theory based on free radical and radiation chemistry. J Gerontol. 1956 Jul;11(3):298-300. doi: 10.1093/geronj/11.3.298. No abstract available. PMID 13332224
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Lee SA, Sypniewski C, Bensadon BA, McLaren C, Donahoo WT, Sibille KT, Anton S. Determinants of Adherence in Time-Restricted Feeding in Older Adults: Lessons from a Pilot Study. Nutrients. 2020 Mar 24;12(3):874. doi: 10.3390/nu12030874. PMID 32213965
- [Background] Martens CR, Rossman MJ, Mazzo MR, Jankowski LR, Nagy EE, Denman BA, Richey JJ, Johnson SA, Ziemba BP, Wang Y, Peterson CM, Chonchol M, Seals DR. Short-term time-restricted feeding is safe and feasible in non-obese healthy midlife and older adults. Geroscience. 2020 Apr;42(2):667-686. doi: 10.1007/s11357-020-00156-6. Epub 2020 Jan 23. PMID 31975053
- [Background] Mattson MP, Moehl K, Ghena N, Schmaedick M, Cheng A. Intermittent metabolic switching, neuroplasticity and brain health. Nat Rev Neurosci. 2018 Feb;19(2):63-80. doi: 10.1038/nrn.2017.156. Epub 2018 Jan 11. PMID 29321682
- [Background] McCay CM, Crowell MF, Maynard LA. The effect of retarded growth upon the length of life span and upon the ultimate body size. 1935. Nutrition. 1989 May-Jun;5(3):155-71; discussion 172. No abstract available. PMID 2520283
- [Background] Mitchell SJ, Bernier M, Mattison JA, Aon MA, Kaiser TA, Anson RM, Ikeno Y, Anderson RM, Ingram DK, de Cabo R. Daily Fasting Improves Health and Survival in Male Mice Independent of Diet Composition and Calories. Cell Metab. 2019 Jan 8;29(1):221-228.e3. doi: 10.1016/j.cmet.2018.08.011. Epub 2018 Sep 6. PMID 30197301
- [Background] Ooi TC, Meramat A, Rajab NF, Shahar S, Ismail IS, Azam AA, Sharif R. Intermittent Fasting Enhanced the Cognitive Function in Older Adults with Mild Cognitive Impairment by Inducing Biochemical and Metabolic changes: A 3-Year Progressive Study. Nutrients. 2020 Aug 30;12(9):2644. doi: 10.3390/nu12092644. PMID 32872655
- [Background] Ooi TC, Meramat A, Rajab NF, Shahar S, Sharif R. Antioxidant Potential, DNA Damage, Inflammation, Glycemic Control and Lipid Metabolism Alteration: A Mediation Analysis of Islamic Sunnah Intermittent Fasting on Cognitive Function among Older Adults with Mild Cognitive Impairment. J Nutr Health Aging. 2022;26(3):272-281. doi: 10.1007/s12603-022-1757-0. PMID 35297471
- [Background] Reiman EM, Caselli RJ, Yun LS, Chen K, Bandy D, Minoshima S, Thibodeau SN, Osborne D. Preclinical evidence of Alzheimer's disease in persons homozygous for the epsilon 4 allele for apolipoprotein E. N Engl J Med. 1996 Mar 21;334(12):752-8. doi: 10.1056/NEJM199603213341202. PMID 8592548
- [Background] Rey, A. (1964). L'examen clinique en psychologie. Paris, Presses Universitaires de France.
- [Background] Reynolds, C. R. (2002). Comprehensive trail-making test : examiner's manual. Austin, Tex., Pro-Ed.
- [Background] Roy M, Rheault F, Croteau E, Castellano CA, Fortier M, St-Pierre V, Houde JC, Turcotte EE, Bocti C, Fulop T, Cunnane SC, Descoteaux M. Fascicle- and Glucose-Specific Deterioration in White Matter Energy Supply in Alzheimer's Disease. J Alzheimers Dis. 2020;76(3):863-881. doi: 10.3233/JAD-200213. PMID 32568202
- [Background] Rubinsztein DC, Frake RA. Yoshinori Ohsumi's Nobel Prize for mechanisms of autophagy: from basic yeast biology to therapeutic potential. J R Coll Physicians Edinb. 2016 Dec;46(4):228-233. doi: 10.4997/jrcpe.2016.403. PMID 28504774
- [Background] Sattler MC, Jaunig J, Tosch C, Watson ED, Mokkink LB, Dietz P, van Poppel MNM. Current Evidence of Measurement Properties of Physical Activity Questionnaires for Older Adults: An Updated Systematic Review. Sports Med. 2020 Jul;50(7):1271-1315. doi: 10.1007/s40279-020-01268-x. PMID 32125670
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Wechsler, D. (1997). Wechsler Adult Intelligence Scale-III. New York, The Psychological Corporation.
- [Background] Weindruch R. The retardation of aging by caloric restriction: studies in rodents and primates. Toxicol Pathol. 1996 Nov-Dec;24(6):742-5. doi: 10.1177/019262339602400618. PMID 8994305
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Wilson, K. G., Sandoz, E. K., Kitchens, J., & Roberts, M. E. (2010).